CLINICAL TRIAL: NCT03940989
Title: The Impact of Dosing Parameters on Motor Skill Acquisition and Retention in Bilateral Cerebral Palsy (BCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Teachers College, Columbia University (Other)
Responsible Party: Principal Investigator, Susan Sienko, Research Associate, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 79142
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor blinded to activities that the participant is working on during camp
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-Week Camp (Experimental): Subject will participate in a HABIT-ILE camp format for 6-hours/day, 5 days/week for three weeks.
  Interventions: Other: HABIT-ILE
- 15-Week Camp (Experimental): Subject will participate in a HABIT-ILE camp format for 6-hours/day, one day/week for 15 weeks.
  Interventions: Other: HABIT-ILE

INTERVENTIONS:
Other: HABIT-ILE — Goal-directed, task-specific training for both the upper (UE) and lower extremity (LE) and postural control.

SUMMARY:
A recent systematic review found that therapeutic interventions that apply principles of motor learning with intense practice improve functional upper extremity movement in children with unilateral CP. Evidence of efficacy for any treatment approach aimed at improving motor function in bilateral CP (the most prevalent form) is lacking. Preliminary investigation suggests that intensive (90 hours) goal-directed, task-specific training provided in a 3-week day camp format can improve functional movement of both the upper (UE) and lower extremity (LE) and postural control in children with BCP. To date, HABIT-ILE has only been provided in a day camp setting over several weeks. Implementing the dosing schedule of this promising intensive approach in a hospital setting requires innovative resource allocation (space and staff); thus, examining alternative delivery models is imperative. The purpose of this study is to conduct a multi-center randomized control trial (RCT) to determine whether 90 hours of HABIT-ILE improves functional motor skills, activity and motivation in children with BCP when dosed in a camp format at 6-hours/day, 5 days/week for three weeks and 6-hours/day, one day/week for 15 weeks.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the leading cause of childhood motor impairment with 1 in 323 American children affected. The resulting impaired motor function in individuals with CP limits their ability to independently perform many functional activities, and participate in academic, social, and leisure activities. Children with CP are referred to physical, occupational, and speech therapy at varying intensities (1-3x week) for years, depending on individual needs. While these therapeutic services are offered regularly, the clinical efficacy and optimal dosing parameters are being challenged. In a meta-analysis of all available therapeutic interventions for CP, just 5 had strong enough evidence to recommend implementation into clinical practice for children with unilateral CP (Novak et al. 2013) and no therapies had sufficient evidence of efficacy for treatment of upper (UE) or lower extremities (LE) in children with bilateral CP (BCP). The key features of interventions with proven evidence of clinical efficacy include: a motor learning approach involving active movement, an environment to shape desired movements, and a much higher treatment intensity than provided in weekly therapies. Despite BCP being the most prevalent subtype, the majority of the research evaluating the clinical efficacy and dosing parameters of therapeutic interventions has been determined in children with UCP with upper extremity approaches such as Constraint Induced Movement Therapy (CIMT) and Hand-Arm Bimanual Intensive Therapy (HABIT) demonstrating efficacy.

One promising therapy gaining interest and support for children with BCP is Hand-Arm Bimanual Intensive Therapy Including the Lower Extremities (HABIT-ILE). HABIT-ILE aims to improve upper and lower movement control by engaging the UE and LE during combined activities for many hours every day for 3 weeks. Preliminary investigation has demonstrated that children with BCP participating in a 90-hour HABIT-ILE day camp achieve improvement within the body function and structure, activity and participation levels of the International Classification of Functioning, Disability and Health (ICF). While intensive therapies, such as HABIT-ILE, are typically provided in a day camp setting over several weeks, implementing the dosing schedule of this promising intensive approach in a hospital setting requires innovative resource allocation (space and staff). In order to establish the efficacy of this approach for children with BCP, it is essential to further examine the efficacy of the 3-week HABIT-ILE camp format of delivery in a larger, multisite trial, in addition to examining whether an alternative model of intensity and resource allocation can demonstrate similar efficacy. The overall aim of the proposed work is to determine the effectiveness of two different dosing schedules of an intensive therapeutic intervention that applies motor learning to upper and lower extremity movement and postural control to improve functional motor skills, activity, and self-mastery in children with BCP. The specific aims are:

Specific Aim 1: To determine if there are significant gains and retention in functional motor skills, activity, and self-mastery in children with BCP receiving 90 hours of HABIT-ILE dosed in a camp format for 6-hours per day, 5 days per week for three weeks and for 6-hours a day, one day per week for 15 weeks.

Specific Aim 2: To determine whether the degree of involvement, age and self-mastery predict the magnitude and maintenance of change seen in children with BCP receiving 90 hours of HABIT-ILE dosed in a camp format for 6-hours per day, 5 days per week for three weeks and for 6-hours a day, one day per week for 15 weeks.

ELIGIBILITY:
Need to live within commuting distance of Columbia University (NY, NY), Shriners Hospitals for Children-Greenville (Greenville, SC) or Shriners Hospitals for Children-Portland (Portland, OR)

Inclusion Criteria:

* Diagnosis of Bilateral Cerebral Palsy
* Gross Motor Function Classification System (GMFCS) levels II-IV
* Able to get up from a chair with standby assist
* Able to sit on a mat table with upper extremity support
* Ability to understand directions
* Ability to walk 10 steps with/without assistive device and standby assist
* Ability to understand and speak english
* Willing to restrict Botox/Dysport use for 3 months prior to each of the 4 full assessments
* Willing to be randomized to either camp format

Exclusion Criteria:

* Traumatic Brain Injury
* Predominate Dystonia
* Predominate Athetosis
* Orthopedic surgery in the last year or plans during the study period

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure (GMFM) | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  Objective assessment of crawling, kneeling, standing, walking, running, jumping.The GMFM is scored on a 4-point scale ranging from does not initiate (0) to completes (3). Each dimension is scored independently providing a measure of functional motor ability within the dimension.
Change in Jebsen-Taylor Test of Hand Function | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  Objective test of hand function for activities of daily living. Scoring is based on time to perform the individual tasks and times are compared to normative tables with assessment by age and gender.
Change in Pediatric Balance Scale | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  Assessment of Standing Balance. THE PBS is a 14 item performance based balance test which is scored on a 5-point scale ranging from a low of 0 to a maximum of 4, with a maximum score of 56.
Change in Trunk Control Measurement Scale | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  The TCMS assesses trunk control during both static and dynamic sitting balance. Dynamic sitting is further divided into selective movement control and dynamic reaching. Higher scores indicate greater balance.

SECONDARY OUTCOMES:
Change in Box and Blocks | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  Grasping, transporting and releasing blocks. The test is performed three times for each hand and the mean number of blocks transferred in a minute from the trials will be used to assess gains in manual dexterity.
Change in 2-minute walk | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  The total distance walked in 2 minutes will be used to assess changes in mobility.
Change in ABILOCO | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  The ABILOCO-kids is a 10-item parent-report measure of locomotor ability for children with lower limb impairments. The items represent continuous progression in difficulty of the locomotor activity.
Change in ABILHAND | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  The ABILHAND-kids is a 21-item parent-report measure of bimanual activity for children with CP. The bimanual activities demonstrate continuous progression in difficulty. Higher scores indicate greater ability.
Change in Pediatric Evaluation of Disability Inventory (PEDI-CAT) | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  Parent questionnaire to assess both capability and performance of functional activities in self-care, mobility, and social function. Each of the three scales will be assessed separately to determine whether specific functional activity areas change with intervention. Higher scores indicate a higher functional level.
Change in Dimensions of Mastery Questionnaire | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  The 45-item parent-report questionnaire assesses two elements of mastery motivation: instrumental (persistence at object-related tasks, social activities with adults, social interactions with peers, and gross motor tasks) and expressive (behavioral indicators of positive affect during or following tasks and negative reaction to failure). Subscale scores will be used to determine whether motivation impacts gains in functional motor skills and whether gains in functional motor skills impact the magnitude of motivation.
Change in Canadian Occupational Performance Measure (COPM) | One assessment at Baseline will be used to define goals. Two end of study evaluations (EOS) one the week after completion of camp and a 6-month followup
  Semi-structured interview that enables and open dialogue between the patient/parent on issues of importance to the patient/parent. The COPM is an individualized measure designed to detect change in a child's self-reported occupational performance over time. Occupations are classified into three categories: self-care, productivity and leisure.
Change in Functional and quantitative muscle strength | 3 Assessments: Baseline will be just before the start of camp. Two end of study evaluations: one the week following completion of camp and one at 6-months followup
  Measurement of muscle strength.Quantitative strength of the abductors, knee extensors, and ankle plantarflexors will be measured with a hand-held dynamometer. Functional assessments of standing heel rise, sit to stand and lateral steps ups will assess functional strength. Higher numbers indicate greater strength.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sienko, PhD, Principal Investigator — Shriners Hospitals for Children-Portland
Locations (2):
- United States (2):
  - Teachers College, Columbia University, New York, New York
  - Shriners Hospitals for Children, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No